CLINICAL TRIAL: NCT04842266
Title: A Prospective Study of the IlluminOss Photodynamic Bone Stabilization System for the Treatment of Impending and Actual Pathological Fractures in the Pelvis From Metastatic Bone Disease or Geriatric Pelvic Fractures
Brief Title: IlluminOss Photodynamic Bone Stabilization System for the Treatment of Impending and Actual Pelvis Fractures
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: IlluminOss Medical, Inc. (Industry); University of Miami (Other)
Responsible Party: Principal Investigator, Kevin A.Raskin, MD, Physician, Massachusetts General Hospital
Other Study IDs: 2021P000047
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cancer Metastatic; Trauma; Pathologic Fracture
MeSH Terms: conditions — Neoplasm Metastasis; Wounds and Injuries; Fractures, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Impending or actual non-displaced or minimally displaced pathologic fractures of the pelvis: Patients are being targeted because they have already agreed to the undergo the IlluminOss Pelvic Implant for standard clinical care. Patient-reported outcome surveys will be administered pre-operatively, as well as at 2 days, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years after surgery.
  Interventions: Device: IlluminOss pelvic implant for oncologic indication
- Pelvic fragility fracture in a geriatric patients (age 65 or older): Patients are being targeted because they have already agreed to the undergo the IlluminOss Pelvic Implant for standard clinical care. Patient-reported outcome surveys will be administered pre-operatively, as well as at 2 days, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years after surgery.
  Interventions: Device: IlluminOss pelvic implant for geriatric trauma indication

INTERVENTIONS:
Device: IlluminOss pelvic implant for oncologic indication — Impending or actual non-displaced or minimally displaced pathologic fractures of the pelvis
  Groups: Impending or actual non-displaced or minimally displaced pathologic fractures of the pelvis
Device: IlluminOss pelvic implant for geriatric trauma indication — Pelvic fragility fracture in a geriatric patients (age 65 or older)
  Groups: Pelvic fragility fracture in a geriatric patients (age 65 or older)

SUMMARY:
The aim of this project is to assess the effectiveness of the IlluminOss pelvic implants in patients with pelvic metastatic disease presenting with pain, risk of pathologic fracture, non-displaced or minimally displaced pathologic fracture of the pelvis, and geriatric patients with pelvic fragility fractures. Results from this study will be used to confirm preliminary clinically and possibly statistically significant reductions in pain and improvements in function among these patients.

DETAILED DESCRIPTION:
The matrix morphology of the tumors in metastatic bone disease (MBD) may be of blastic, lytic, or mixed characteristics. Cancers of purely lytic or mixed blastic-lytic composition are the most concerning, as they result in local destruction of the cortical and trabecular bone, causing significant pain and increasing the risk of a pathologic fracture. Function and mobility are severely affected in this patient population due to mechanical and oncogenic pain.

Prophylactic fixation of impending pathological fractures from MBD has demonstrated significant clinical benefit in terms of reducing mechanical pain and in decreasing the progression to complete pathologic fracture as well as minimizing the symptoms when these occur. In the later clinical scenario, the degree of fracture displacement, pain and functional limitation in most cases is minimal as the fracture is an already treated condition. In terms of surgical impact to the patient, prophylactic fixation is a faster procedure with lower blood loss rates. Other benefits include, shorter length of hospitalization and higher likelihood of discharge to home, in addition to reduction of pain, improvement in activities of daily living, and better quality of life.

Importantly, efforts have been made to predict fracture risk and the need for prophylactic fixation based upon the clinical and radiographic features of MBD. This is well stablished in long bones of the extremities but it is not as clear or conclusive in the pelvis.

Traditionally, Intramedullary devices are used for the purposes of prophylactic fixation and for treatment of pathologic fractures. Advantages include protection of the whole bone and ability to early bear weight given the biomechanical characteristics as a load sharing device. More commonly, these implants are made of titanium or other metal alloys. In recent years, the development of radiolucent implants has been important in orthopaedic oncology as these facilitate evaluation of bone involvement and radiation therapy planning. One of these radiolucent devices is IlluminOss PBSS. This UV light activated polymer has proved to be effective and safe in the treatment of impending pathologic fractures of the humerus. This intramedullary implant is inserted through small incisions and proved to be as effective as traditional intramedullary nails in relieving pain and returning patients faster to their pre-impending fracture level of activity. This product has been cleared by the FDA for use in the humerus, radius and ulna, clavicle, pelvis, fibula, metacarpals, metatarsals, and phalanges. The IlluminOss Photodynamic Bone Stabilization System can also be used in conjunction with FDA-cleared fracture fixation systems to provide supplemental fixation in these anatomic sites. The IlluminOss System may be used in the femur and tibia to provide supplemental fixation to an anatomically appropriate FDA-cleared fracture fixation system.

Pelvic fractures in the elderly are a growing concern as the population ages. While oftentimes treated non-operatively, some require surgical fixation. In addition to the stress which surgery especially puts on geriatric patients, a return to pre-injury mobility is also an important impact and a concern of such procedures.

Contrary to the extremities, there are minimal options for small incision pelvic implants to treat patients suffering from pain or fracture. The complex anatomy of the pelvis does not allow the use of rigid and precontoured implants. Fixation with screws is also challenging given the complex anatomy and high prevalence of vital neurovascular structures in the pelvis.

The non-rigid nature of this polymer in the IlluminOss PBSS makes it suitable to adapt to the complex anatomy of the pelvis. In addition, there is no need to use screws for additional fixation, which is ideal in the pelvis. This implant may allow surgeons to forego the use of screws for fixation because the implant has a 3D anti-rotational profile which generates intrinsic stability when in contact with the inner bone. However, if the surgeon considers that stability is not sufficient, screws may still be used in this study at the surgeon's discretion.

This device has been approved to be used in the pelvis after the experience in a previous study examining its effectiveness in the humerus, radius, and ulna. The purpose of this study is to collect information to effectively measure the improvement in pain control through functional scores after the surgery. We wish to see short term results (2 years) and to have a better understanding of the complication profile.

ELIGIBILITY:
Inclusion criteria:

Patients are being targeted because they have already agreed to the undergo the IlluminOss Pelvic Implant for standard clinical care. It is a decision made by the treating surgeon separately from research and prior to mention of the study.

1. Patient is a skeletally mature patient 21 years of age or older (closed epiphyseal plates) who receiving the FDA-approved IlluminOss Pelvic Implant
2. IlluminOss Pelvic Implant is intended to treat pain due to impending or actual non-displaced or minimally displaced pathologic fractures of the pelvis secondary to metastatic malignancy, multiple myeloma, lymphoma, or radiation osteitis or a pelvic fragility fracture in a geriatric patients (age 65 or older)
3. VAS Pain Score ≥ 30 on 0 to 100 scale

Exclusion criteria:

1. Patient is uncooperative, or patient incapable of following directions (for example, as a consequence of a neurological or psychiatric disorder)
2. Patient is a prisoner
3. Patient is deemed surgically unfit by the medical oncology service

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skeletally mature patients with undergoing surgery to treat pain due to impending or actual non-displaced or minimally displaced pathologic fractures of the pelvis secondary to metastatic malignancy, multiple myeloma, lymphoma, or radiation osteitis or a pelvic fragility fracture in a geriatric patients (age 65 or older).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survey of patient-reported outcomes | Pre-operatively through 2 years after surgery
  Patients treated with the IlluminOss pelvic implant will be given functional and pain surveys pre-operatively (within 2 weeks before surgery) and post-operatively (at 2 days, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years). 100 patients will be included in the study. The surveys include the VAS Pain, the EQ-VAS, the Combined Pain and Ambulatory Function, the PROMIS Pain Inteference, and the PROMIS Physical Function. Additionally, the MSTS survey will be collected for oncologic patients. If needed, the surveys will be mailed to the patient with a pre-stamped and pre-addressed envelope. When mailing patients MSTS surveys, we will include a set of instructions to guide participants through the questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gausepohl T, Pennig D, Heck S, Gick S, Vegt PA, Block JE. Effective Management of Bone Fractures with the Illuminoss(R) Photodynamic Bone Stabilization System: Initial Clinical Experience from the European Union Registry. Orthop Rev (Pavia). 2017 Feb 20;9(1):6988. doi: 10.4081/or.2017.6988. eCollection 2017 Feb 20. PMID 28286623
- [Background] Surke C, Meier R, Haug L, Vogelin E. Osteosynthesis of fifth metacarpal neck fractures with a photodynamic polymer bone stabilization system. J Hand Surg Eur Vol. 2020 Feb;45(2):119-125. doi: 10.1177/1753193419880775. Epub 2019 Oct 22. PMID 31635518
- [Background] Van Oijen GW, Vegt PA, Hagenaars T, Van Lieshout EMM, Verhofstad MHJ. Outcome after treatment of distal radius fractures in the elderly using the IlluminOss(R) System. Eur J Trauma Emerg Surg. 2021 Aug;47(4):1129-1136. doi: 10.1007/s00068-019-01289-w. Epub 2020 Jan 16. PMID 31950234
- [Background] Vegt P, Muir JM, Block JE. The Photodynamic Bone Stabilization System: a minimally invasive, percutaneous intramedullary polymeric osteosynthesis for simple and complex long bone fractures. Med Devices (Auckl). 2014 Dec 12;7:453-61. doi: 10.2147/MDER.S71790. eCollection 2014. PMID 25540600
- [Background] Stumpf M, Kraus T, Plotz W, Jakobs TF. [Stabilization of the pelvic ring with photodynamic bone stabilization (IlluminOss)]. Unfallchirurg. 2015 Mar;118(3):279-82. doi: 10.1007/s00113-015-2743-3. German. PMID 25783693
- [Background] Hagenaars T, Van Oijen GW, Roerdink WH, Vegt PA, Vroemen JP, Verhofstad MH, Van Lieshout EM. Functional recovery after treatment of extra-articular distal radius fractures in the elderly using the IlluminOss(R) System (IO-Wrist); a multicenter prospective observational study. BMC Musculoskelet Disord. 2016 May 27;17:235. doi: 10.1186/s12891-016-1077-9. PMID 27233355
- [Background] Zyskowski M, Cronlein M, Heidt E, Biberthaler P, Kirchhoff C. [Osteosynthesis of distal fibular fractures with IlluminOss : Video article]. Unfallchirurg. 2017 Jan;120(1):6-11. doi: 10.1007/s00113-016-0285-y. German. PMID 27987018